CLINICAL TRIAL: NCT02615743
Title: Automated Adherence Feedback for High Risk Children With Asthma
Brief Title: Asthma Controller Adherence After Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-012092
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Caregivers of intervention arm participants will receive daily text message reminders about asthma controller medication use, as well as an electronic monitoring device to track the participant's medication usage for 60 days following hospital discharge. At the end of 30 days, participants will be able to opt out of daily text messages if they choose. All caregivers of participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  Interventions: Behavioral: Daily Text message reminder; Device: Inhaled steroid canister monitor
- Control Group (Other): Caregivers of control arm participants will receive an electronic monitoring device to track their medication usage for 60 days following hospital discharge. At 30 days, caregivers of participants will be able to opt in to receive daily text message reminders about asthma medication use. Caregivers of all participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  Interventions: Device: Inhaled steroid canister monitor

INTERVENTIONS:
Behavioral: Daily Text message reminder — Subjects in the intervention arm will receive once daily text messages at the time of their choice or at a default time of 7am. The text message will remind them to give their child their controller medication and provide a helpful information on asthma controller use.
  Arms: Intervention Group
Device: Inhaled steroid canister monitor — An electronic monitor will be affixed to subjects' inhaled steroid canister and families will be instructed to use the inhaler as directed by their physician. Subjects will not receive daily text messages.The canister monitor, the Propeller sensor (Propeller, Madison, Wisconsin) is an FDA-approved, portable device which affixes to the top of most metered dose inhaler canisters. The devices records the number and time of each inhaler actuation and transmits this information to either a smart phone or cellular modem. Data is then sent via the cellular network to the secure Propeller server. The data will then be downloaded monthly.
  Other Names: Propeller Health Bluetooth Low Energy (BLE) Sensor

SUMMARY:
This study sets out to assess whether daily text message reminders help to enhance the consistency of use of controller medications following hospitalization for pediatric asthma patients ages 4-11 and their families. Text message reminders will be delivered to a subject's cell phone for those in the intervention group and electronic monitors will placed on the controller inhalers at the time of hospital discharge to track medication use over time in both the intervention and the regular care group. Families will complete surveys on the day of enrollment (in person), day 30 (telephone) and day 60 (telephone) on aspects of asthma care including asthma knowledge, medication routines, who is responsible for asthma care, and medication beliefs.

DETAILED DESCRIPTION:
Poor adherence to inhaled controller medications for asthma is a well-documented and poorly understood problem with a disproportionate prevalence and impact on urban minority children. Recent randomized trials from other countries using electronic monitoring of inhaled steroids with automated adherence feedback demonstrated dramatic improvements in adherence behavior. Whether similar intervention effects can be expected in high-risk children in the US is unknown.

To accomplish the above objectives, investigators propose to enroll 40 children and their parents (20 parent/child dyads in each arm) in a two-month pilot randomized controlled trial of an automated adherence feedback intervention. Children will be from West Philadelphia, ages 4-11, and must be hospitalized for asthma at The Children's Hospital of Philadelphia (CHOP).

The study intervention will include daily automated medication reminders via text messaging for those subjects randomized to the intervention group. Inhaled controller medication adherence will be measured in both groups using electronic monitors affixed to the top of the canister of the inhaled steroid medication and adherence trajectories will be determined using group-based trajectory modeling. Factors associated with adherence trajectories will be assessed using a survey completed upon enrollment, completion of the treatment phase (1 month) and upon completion of follow up (2 months). Feasibility outcomes will include use, acceptance, and preferences. Limited efficacy outcomes will include change in parent-reported asthma control and difference in average percent adherence between intervention and control conditions.

Findings from this study will provide preliminary data for a larger study evaluating the mechanisms of differential adherence trajectories and the effect of an adherence feedback intervention for different mechanisms of non-adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Has unlimited text messaging plan
2. Prescribed one of the following metered dose inhalers for daily use: Flovent (fluticasone), QVAR (budesonide), Seretide (fluticasone-salmeterol), Advair multi-dose inhaler (MDI) (fluticasone-salmeterol) or Dulera (mometasone-formoterol)
3. Patient receives primary care at one of the three urban CHOP primary care practices (Karabots, South Philadelphia, and Cobbs Creek)

Exclusion Criteria:

1. Subjects prescribed a controller medication to which the electronic device cannot affix (i.e. montelukast, Advair Diskus, Symbicort, Seretide Acuhaler/Diskus) as their primary controller medication
2. Subjects with developmental delays or disabilities
3. Families with active Department of Human Services (DHS) involvement
4. Non-English speaking families
5. Parents/guardians or subjects who the inpatient medical team recommends against approaching for enrollment in a research study

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09-20 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen C Kenyon, MD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Adams SA, Leach MC, Feudtner C, Miller VA, Kenyon CC. Automated Adherence Reminders for High Risk Children With Asthma: A Research Protocol. JMIR Res Protoc. 2017 Mar 27;6(3):e48. doi: 10.2196/resprot.6674. PMID 28347975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children were the participants enrolled in the study, parents/caregivers were not.
Groups:
- Intervention Group: Caregivers of Intervention arm participants will receive daily text message reminders about asthma controller medication use, as well as an electronic monitoring device to track their medication usage for 60 days following hospital discharge. All participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  The text message will remind them to give their child their controller medication and provide a helpful information on asthma controller use.
  An electronic monitor will be affixed to subjects' inhaled steroid canister and families will be instructed to use the inhaler as directed by their physician. The canister monitor, the Propeller sensor (Propeller, Madison, Wisconsin) is an FDA-approved, portable device which affixes to the top of most metered dose inhaler canisters. The devices records the number and time of each inhaler actuation and transmits this information to either a smart phone or cellular modem.
- Control Group: Caregivers of control arm participants will receive an electronic monitoring device to track their medication usage for 60 days following hospital discharge. All participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  An electronic monitor will be affixed to subjects' inhaled steroid canister and families will be instructed to use the inhaler as directed by their physician. Subjects will not receive daily text messages.The canister monitor, the Propeller sensor (Propeller, Madison, Wisconsin) is an FDA-approved, portable device which affixes to the top of most metered dose inhaler canisters. The devices records the number and time of each inhaler actuation and transmits this information to either a smart phone or cellular modem.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 21 | 20
Completed | 15 | 17
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Caregivers of intervention participants will receive daily text message reminders about asthma controller medication use and an electronic monitoring device to track their medication use for 60 days following hospital discharge. All caregivers of participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  The text message will remind them to give their child their controller medication and provide a helpful information on asthma controller use.
  An electronic monitor will be affixed to subjects' inhaled steroid canister and families will be instructed to use the inhaler as directed by their physician. The canister monitor, the Propeller sensor (Propeller, Madison, Wisconsin) is an FDA-approved, portable device which affixes to the top of most metered dose inhaler canisters. The devices records the number and time of each inhaler actuation and transmits this information to either a smart phone or cellular modem.
- Control Group: Caregivers of control arm participants will receive an electronic monitoring device to track their medication usage for 60 days following hospital discharge. All caregivers of participants will also complete a 30-minute survey at the time of enrollment and 2 brief telephone followups at 30 and 60 days.
  An electronic monitor will be affixed to subjects' inhaled steroid canister and families will be instructed to use the inhaler as directed by their physician. Subjects will not receive daily text messages.The canister monitor, the Propeller sensor (Propeller, Madison, Wisconsin) is an FDA-approved, portable device which affixes to the top of most metered dose inhaler canisters. The devices records the number and time of each inhaler actuation and transmits this information to either a smart phone or cellular modem.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (2.1) | 5.8 (2.1) | 5.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 20 | 15 | 35
  Other | 1 | 5 | 6
Primary Caregiver Education [Number; unit: primary caregiver of participant]
  High School or less | 14 | 7 | 21
  Some College and above | 7 | 13 | 20
Family Income Level [Count of Participants; unit: Participants]
  <$30,000 | 15 | 12 | 27
  >$30,000 | 6 | 8 | 14
Child Health Insurance [Count of Participants; unit: Participants]
  private | 1 | 4 | 5
  public | 20 | 16 | 36
Baseline Caregiver Asthma Knowledge Questionnaire [Mean (Standard Deviation); unit: percentage score] — The minimum score is a 0 and the maximum is 100. Higher values are better scores meaning better Asthma knowledge.
  percentage score | 93 (8.7) | 92 (8.4) | 93 (8.5)
Baseline child Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — Asthma Control Test (ACT) provides a numerical score to determine if asthma symptoms are well controlled. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well controlled asthma.
  units on a scale | 17.8 (4.3) | 17.2 (4.7) | 17.3 (4.4)
Baseline prior adherence (caregiver-reported), mean (std) [Mean (Standard Deviation); unit: percentage of medication taken] — Participants indicate, on a scale of 0-10, how much controller medication their child took in the last month. 10 means they took every single dose of medication (100%), 5 means half, and 0 means that their child took no medication.
  percentage of medication taken | 65 (23) | 62 (25) | 64 (24)
Baseline adherence intent , mean (std) [Mean (Standard Deviation); unit: percentage of intended medication] — Participants indicate, on a scale of 0-10, how much controller medication their child will take in the next month. 10 means they intend to take every single dose of medication (100%), 5 means half, and 0 means that they intend to not take any medication.
  percentage of intended medication | 80 (23) | 85 (21) | 85 (21)
Prior asthma-related emergency department visits in year before enrollment, mean (std) [Mean (Standard Deviation); unit: visits] | 1.0 (1.5) | 1.0 (1.6) | 1.0 (1.5)
Prior asthma-related hospitalizations in year before enrollment, mean (std) [Mean (Standard Deviation); unit: hospitalizations] | 0.3 (0.6) | 0.5 (0.8) | 0.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Number and Percentage of Patients That Use Monitoring Device Over 30 Days (Feasibility)
Description: The number and percentage of patients that continue to use the monitoring device throughout the month will be compared between the intervention and control groups.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 21 | 20
Participants | 15 | 17

2. Primary Outcome: Acceptability
Description: The rating of the monitoring device will be compared between groups based on responses to a questionnaire asking about acceptability and preferences to determine if there is a difference in the "favorability" We determined this by the number of participants who found text message reminders helpful to avoid missing doses. After 30 days caregivers of control group participants were given the option to receive daily text messages; they were asked about acceptability 30 days later.
Time Frame: 30 days (intervention group) 60 days (control group)
Population: There were 6 participants missing from the intervention group due to loss to followup. There were only 5 caregivers of participants in the control group who agreed to receive daily text messages.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 5
Participants | 15 | 5

3. Secondary Outcome: Adherence
Description: Percent adherence will be calculated as observed medication actuations from electronic adherence monitors over expected use (the latter is = prescribed daily regimen number of observation days)
Time Frame: 30 days
Population: There are only 15 participants in the intervention group and 17 in the control group due to loss to follow up.
Measure: Mean (95% Confidence Interval); unit: percent adherence
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 17
percent adherence | 34 [18 to 50] | 40 [25 to 55]

4. Secondary Outcome: Change in Child Asthma Control Tool Score (cACT) From Baseline to End of Intervention Period.
Description: The difference in the change of cACT score from first study visit to the third study visit will be compared between the two study groups. Asthma Control Test (ACT) provides a numerical score to determine if asthma symptoms are well controlled. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well controlled asthma.
Time Frame: 30 days
Population: There are only 15 participants in the intervention group and 17 in the control group due to loss to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 17
units on a scale | 1.0 (2.8) | 3.1 (3.0)

ADVERSE EVENTS:
Time Frame: 60 days
Description: No adverse events, serious or other, were reported during by any participants during this pilot study.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No